CLINICAL TRIAL: NCT07240610
Title: Observational Study on the Abscopal Efect by Ultra-hypofractionated Radiation Therapyin Combination With Immune Checkpoint Inhibiters for Metastatic Renal Cell Carcinoma
Brief Title: Abscopal Effect of Ultra-Hypofractionated Radiation Plus Immunotherapy in Metastatic Renal Cell Carcinoma
Acronym: AURICRE
Status: Recruiting | Type: Observational
Sponsor: Zhe Chen (Other)
Collaborators: Participating institutions of the AURICRE Study Group (Unknown)
Responsible Party: Sponsor-Investigator, Zhe Chen, Lecturer, University of Yamanashi
Organization: University of Yamanashi (Other)
Other Study IDs: CS0075; UMIN000059652 (Other: University Hospital Medical Information Network (UMIN)); JP24K02397 (Other: Japan Society for the Promotion of Science (JSPS))
Record Dates: First submitted 2025-11-16; First posted 2025-11-21 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Renal Cell Cancer Metastatic
Keywords: Abscopal Effect; Ultra-Hypofractionated Radiotherapy; Immune Checkpoint Inhibitors; Metastatic Renal Cell Carcinoma; Immunoradiotherapy Combination
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Peripheral blood samples (serum and plasma) for cytokine analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mRCC patients receiving ICIs and IGU: This cohort includes patients with histologically confirmed mRCC who are receiving ICIs and undergo IGU to a selected metastatic lesion as part of their standard clinical care. Patients are followed prospectively for one year to evaluate abscopal responses, survival outcomes, and immune-related biomarkers.

SUMMARY:
The goal of this multicenter observational study is to elucidate the clinical and immunological characteristics of the abscopal effect in patients with metastatic renal cell carcinoma (mRCC) receiving immune checkpoint inhibitors (ICI) combined with image-guided ultra-hypofractionated radiotherapy (IGU).

The main questions this study aims to answer are:

What is the abscopal response rate (ARR) at one year after IGU in patients continuing ICI treatment?

What clinical and immunological factors are associated with the occurrence and timing of the abscopal effect?

Participants are patients with mRCC who have experienced immune-confirmed stable or progressive disease during ICI therapy and are scheduled to receive IGU to a selected lesion. Researchers will observe tumor responses at irradiated and non-irradiated sites using standard imaging (CT/MRI) and collect clinical and laboratory data at baseline, 3, 6, 9, and 12 months after IGU. Optional exploratory blood samples will be obtained for cytokine analysis (e.g., IFN-β, IFN-γ, TNF-α, IL-6).

The primary outcome is the abscopal response rate (ARR) at one year after IGU. Secondary outcomes include tumor shrinkage rate of irradiated and non-irradiated lesions, 1-year overall survival, disease-specific survival, and progression-free survival.

This study seeks to establish a foundation for developing combined immunotherapy and ultra-hypofractionated radiotherapy strategies for metastatic renal cell carcinoma.

*This study is led by Prof. Hiroshi Onishi (University of Yamanashi). The registry entry is managed by Dr. Zhe Chen on behalf of the study group.

DETAILED DESCRIPTION:
Renal cell carcinoma (RCC) is a highly immunogenic tumor that exhibits intrinsic resistance to cytotoxic chemotherapy and conventional radiotherapy. With the introduction of immune checkpoint inhibitors (ICIs), such as nivolumab and ipilimumab, the survival outcomes of patients with metastatic RCC (mRCC) have markedly improved. However, disease control remains suboptimal in a considerable fraction of patients who experience immune-confirmed stable disease or progression despite continued ICI therapy. For such patients, locoregional treatment targeting oligoprogressive lesions may modulate tumor immunogenicity and enhance systemic immune responses.

Radiation therapy, particularly when administered in large doses per fraction (ablative or ultra-hypofractionated schedules), can induce systemic antitumor effects mediated by immune activation, known as the abscopal effect. This effect refers to regression of non-irradiated metastatic lesions following local irradiation, thought to arise from radiation-induced antigen release and subsequent immune activation. Although multiple case reports and small series have described this phenomenon, the true frequency, biological basis, and predictive factors of the abscopal effect in mRCC remain poorly defined.

The AURICRE study (Observational Study on the Abscopal Effect by Ultra-Hypofractionated Radiation Therapy in Combination with Immune Checkpoint Inhibitors for Metastatic Renal Cell Carcinoma) is a multicenter prospective observational registry initiated by the Department of Imaging-Integrative Therapeutic Radiology, University of Yamanashi. The study is designed to clarify the incidence, timing, and clinical-immunological correlates of the abscopal effect in patients with mRCC treated with ICIs who undergo ultra-hypofractionated image-guided radiotherapy (IGU) to a metastatic lesion. This investigation will also provide a foundation for the rational development of future ICI-radiotherapy combination strategies.

Study Objectives

Primary Objective To elucidate the clinical and immunological characteristics associated with the abscopal effect in mRCC patients receiving ICIs and to determine the abscopal response rate (ARR) at one year after IGU.

Secondary Objectives

To evaluate:

The tumor shrinkage rate of irradiated and non-irradiated lesions at each follow-up interval

One-year overall survival (OS)

One-year disease-specific survival (DSS)

One-year progression-free survival (PFS)

Exploratory Objectives To explore cytokine dynamics and immune biomarkers (e.g., IFN-β, IFN-γ, TNF-α, IL-6) that may predict or accompany the abscopal effect.

Study Design

This study is a prospective, multicenter, observational design conducted from 2025 to 2028. Eligible patients are adults with histologically confirmed metastatic RCC who have received ICIs and demonstrated immune-confirmed stable disease or progression. Participants must be candidates for ultra-hypofractionated radiotherapy to at least one metastatic lesion according to clinical judgment. There is no randomization or additional therapeutic intervention mandated by the protocol beyond standard care.

Treatment and Assessment Schedule

IGU will be performed using stereotactic or equivalent ultra-hypofractionated techniques (typically 24-30 Gy in 1-3 fractions) targeting a single or limited number of lesions, with attention to organ-at-risk constraints. The selection of the irradiation site and dose prescription will follow institutional standards.

Participants will continue ICI therapy at the discretion of their treating oncologist. Imaging assessments (CT or MRI) will be performed at baseline, and at 3, 6, 9, and 12 months post-IGU to evaluate responses in irradiated and non-irradiated lesions based on RECIST 1.1 criteria and radiological review. Optional exploratory blood sampling for cytokine analysis will be performed at corresponding time points. Clinical status, laboratory parameters, and toxicity will be documented throughout the observation period.

Endpoints and Data Collection

Primary Endpoint

Abscopal response rate (ARR) at one year after IGU, defined as a ≥30 % reduction in the sum of diameters of non-irradiated target lesions without new lesion appearance.

Secondary Endpoints

Tumor shrinkage rates of irradiated and non-irradiated lesions

1-year OS, DSS, and PFS

Patterns and timing of the abscopal response

Exploratory Endpoints

Temporal changes in serum cytokine levels

Correlation between immune parameters and clinical response

Data will be collected using an electronic data capture (EDC) system. Each participating site will record baseline demographics, disease characteristics, treatment details, and follow-up results in standardized formats to ensure uniformity across institutions.

Sample Size and Statistical Considerations

The target accrual is approximately 50-60 patients based on feasibility across participating centers. Statistical analyses will include logistic regression to assess predictors of the abscopal response, incorporating variables such as age, sex, number of lesions, prior lines of therapy, and ICI type. Receiver operating characteristic (ROC) curve analysis will determine optimal cut-off values for significant predictors. Survival outcomes will be estimated using the Kaplan-Meier method. Missing data will be analyzed for pattern and mechanism; if imputation is warranted, multiple imputation or appropriate statistical techniques will be employed.

Ethical Considerations and Oversight

This study is conducted in accordance with the Declaration of Helsinki and the Ethical Guidelines for Medical and Health Research Involving Human Subjects (Japan). The protocol and informed consent documents have been approved by the University of Yamanashi Ethics Committee (approval date: October 27, 2025). Each participating institution will obtain local approval where required. Written informed consent will be obtained from all participants prior to enrollment.

Scientific and Clinical Significance

The AURICRE study will be among the first systematic multicenter efforts to characterize the abscopal effect in mRCC under contemporary immunotherapy settings. By integrating clinical outcomes, radiologic responses, and exploratory immune profiling, this study will clarify real-world frequency and predictors of systemic immune activation triggered by ultra-hypofractionated radiotherapy. The findings are expected to provide a mechanistic and clinical rationale for future prospective trials combining radiotherapy and immunotherapy, ultimately contributing to the advancement of immune-radiotherapeutic strategies for renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years and above with metastatic renal cell carcinoma
2. Patients currently receiving immune checkpoint inhibitor (ICI) therapy who are assessed as having iCPD or iSD according to iRECIST
3. Presence of two or more clinically measurable lesions (assessed by CT, MRI, physical examination, or visual inspection) Note: Osteosclerotic lesions without measurable soft-tissue components are excluded
4. Planned to undergo IGU to the target lesion
5. Provided written informed consent after receiving sufficient explanation of this study Note: Proxy signature is permitted if the patient is physically unable to sign

Exclusion Criteria:

1. Patients with active double cancers (synchronous double cancers or metachronous double cancers with a disease-free interval within 2 years).

   However, carcinoma in situ or intramucosal carcinoma considered cured by treatment, and the following tumors even if within 2 years of disease-free interval are not excluded: gastric cancer stage 0-II (UICC), prostate cancer stage I-III, colorectal cancer stage 0-II, esophageal cancer stage 0-I, breast cancer stage 0-II, endometrial cancer stage I-II, cervical cancer stage 0-II, and thyroid cancer stage I-III. In addition, any cancer with a disease-free interval greater than 2 years is not excluded regardless of stage.
2. Patients with serious comorbidities, such as:

   * severe cardiac disease
   * uncontrolled diabetes mellitus despite continuous insulin therapy
   * myocardial infarction within 6 months
   * uncontrolled hypertension
   * active infections (bacterial, viral, or fungal)
   * diarrhea (watery stool), paralytic ileus, or bowel obstruction
   * autoimmune disease
   * any other severe comorbid condition
3. Patients with clear evidence of idiopathic interstitial pneumonia (usual interstitial pneumonia pattern) on chest X-ray or CT
4. Patients with acute-phase pneumonia
5. Patients with psychiatric disorders or psychiatric symptoms judged to make study participation difficult

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with histologically confirmed metastatic renal cell carcinoma (mRCC) who are receiving ICIs and are candidates for IGU to one or more metastatic lesions. Eligible patients must have immune-confirmed stable disease or progression during ongoing ICI therapy. Enrollment will include patients treated at participating centers of the AURICRE multicenter registry.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Abscopal Response Rate (ARR) at 1 Year After IGU | 12 months after image-guided ultra-hypofractionated radiotherapy (IGU)
  The proportion of patients showing an abscopal response, defined as a ≥30% reduction in the sum of diameters of non-irradiated target lesions without new lesion appearance, evaluated according to RECIST 1.1 criteria. Tumor response will be assessed by radiological imaging (CT or MRI) at each follow-up visit and confirmed by central review.

SECONDARY OUTCOMES:
Tumor Shrinkage Rate of Irradiated and Non-Irradiated Lesions | Baseline to 12 months after IGU
  The percentage change in the sum of diameters of irradiated and non-irradiated lesions from baseline, assessed by RECIST 1.1 at each follow-up (3, 6, 9, and 12 months).
One-Year Overall Survival (OS) | 12 months after IGU
  Overall survival defined as the time from initiation of IGU to death from any cause. Patients alive at the end of follow-up will be censored at the date of last contact.
One-Year Disease-Specific Survival (DSS) | 12 months after IGU
  Disease-specific survival defined as the time from IGU to death due to renal cell carcinoma. Deaths from other causes will be censored at the date of death.
One-Year Progression-Free Survival (PFS) | 12 months after IGU
  Progression-free survival defined as the time from IGU to disease progression or death, whichever occurs first, based on RECIST 1.1 criteria.

OTHER OUTCOMES:
Temporal Changes and Correlation of Serum Cytokine Profiles With Abscopal Response | Baseline to 12 months after IGU
  Quantitative changes in circulating cytokines (IFN-β, IFN-γ, TNF-α, IL-6) measured by enzyme-linked immunosorbent assay (ELISA) at baseline and 3 and 12 months after IGU. Statistical correlations between cytokine dynamics and abscopal response rate will be analyzed using logistic regression and receiver operating characteristic (ROC) analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Onishi, MD, PhD, Principal Investigator — University of Yamanashi
Locations (1):
- University of Yamanashi Hospital, Chūō, Yamanashi, Japan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves identifiable clinical information collected in a multicenter observational registry. Data sharing is restricted by institutional and ethical regulations at participating sites, and access is limited to the study investigators for predefined analyses.